CLINICAL TRIAL: NCT00995228
Title: The Practice of Fluid Management in the Post-anesthetic Care Unit (PACU) in Patients Undergoing Elective Surgery: an Observational Study
Brief Title: Fluid Management in the Post-Anesthetic Care Unit (PACU) at Sourasky Medical Center
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof Idit Matot, director Anesthesiology and intensive care unit, Tel Aviv sourasky medical center
Other Study IDs: TASMC-09-IM-0501-CTIL
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Pulmonary Edema; Acute Lung Injury; Hypertension; Renal Failure
Keywords: overhydration; fluid restriction; post-anesthesia care unit
MeSH Terms: conditions — Pulmonary Edema; Acute Lung Injury; Hypertension; Renal Insufficiency; Water Intoxication

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Peri-operative fluid therapy is a controversial area with few randomized trials to guide practice. Fluid management has a significant influence on outcome following surgery. Yet practically, fluid prescription practice during this period is sub-optimal, resulting in avoidable iatrogenic complications.

Several studies have assessed the effect of a 'liberal' vs. a 'restrictive' perioperative fluid regimen on post-operative outcome. However, most of these studies have focused primarily on intra-operative fluid management, whereas postoperative strategies have been less well defined, even though the immediate postoperative period is of critical importance to the patient's recovery. Moreover, whereas intra-operative fluid administration is monitored by the anesthesiologist, postoperatively it is less supervised and may result in excess or lack of intravenous (IV) fluids. Therefore, fluid management audit at the post-anesthesia care unit (PACU) is of paramount importance for patient healthcare. The objective of this study is to follow and report the current practice of fluid administration in the PACU of Tel Aviv Sourasky Medical Center, for an extended period of time as a first step towards establishing evidence-based guidelines for postoperative fluid management.

DETAILED DESCRIPTION:
Background

Perioperative intravenous (IV) fluid management has been a historically controversial issue in anesthesiology. Accumulating evidence suggest that regulated perioperative fluid management has beneficial effects on postoperative outcomes. A restricted perioperative IV fluid regimen aiming at unchanged body weight resulted in reduced complications after elective colorectal resection (1). In another study, patients receiving a reduced intraoperative fluid volume demonstrated less postoperative complications, lower morbidity rates and shorter hospital stay after intraabdominal surgery (2). Conversely, whereas restricted postoperative IV salt and water intake shortened gastrointestinal (GI) function and hospitalization after colonic resection in one study (3), it had no effect on the same outcomes in another randomized clinical trial (4).

Despite the reported benefits of restrictive fluid therapy, this strategy may be associated with adverse outcomes. Inadequate fluid administration can lead to a reduced effective circulating volume resulting in inefficient tissue perfusion (5-7). On the other hand, overhydration, resulting from perioperative fluid excess, has shown association with deleterious effects on cardiac and pulmonary function (8-12), and on recovery of GI motility (2,3,13), tissue oxygenation (14), wound healing and coagulation (15-16). Erroneous fluid administration is generally associated with increased morbidity and postoperative complications (17-21). Altogether, these observations call for a standardized and regulated fluid therapy throughout the perioperative period taking into account patients' premorbid diseases and type of surgery.

Previous studies have focused primarily on intra-operative fluid management. Postoperative strategies have been less well defined, even though the immediate postoperative period is of critical importance to the patient's recovery. Moreover, whereas intra-operative fluid administration is monitored by the anesthesiologist, postoperatively it is less supervised and may result in excess or lack of IV fluids.

The aim of this study is thus to follow and present the current practice of fluid administration in the PACU of Tel Aviv Sourasky Medical Center, for an extended period of time as a first step towards establishing evidence-based guidelines for postoperative fluid management.

Methods

We will collect data regarding intra- and postoperative fluid administration from the charts of >18 years old ASA I-III patients undergoing elective general or orthopedic surgery. Patients with renal/cardiac failure will be analyzed separately, since their pathology dictates extra caution with fluid therapy. Patients demographics, type of surgery, and the type and volume of fluids given during the operation and PACU stay, will be documented as well as the occurrence of morbidity in PACU, without any interventions. Data collection will be anonymous and will last six months. The setting will be the PACU of the Tal Aviv Sourasky Medical center.

Suggested benefits

The purpose of this data report is to provide an overview on the current practice of fluid management in Tel Aviv Sourasky Medical Center's PACU. We believe that this is a preliminary necessary step towards establishing guidelines for postoperative fluid management.

Study Objective

To describe the contemporary practice of postoperative fluid management in the PACU of the Sourasky Medical Center.

References

1. Brandstrup B, Tonnesen H, Pott F et al (2003). Effects of intravenous fluid restriction on postoperative complications: comparison of two perioperative fluid regimens: a randomized assessor-blinded multicenter trial. Ann Surg 238:641-8.
2. Nisanevich V, Felsenstein I, Matot I, et al (2005). Effect of intraoperative fluid management on outcome after intraabdominal surgery.Anesthesiology.103:25-32.
3. Lobo DN, Bostock KA, Allison SP, et al (2002). Effect of salt and water balance on recovery of gastrointestinal function after elective colonic resection: a randomised controlled trial. Lancet 359:1812-8.
4. MacKay G, Fearon K, O'Dwyer PJ et al (2006). Randomized clinical trial of the effect of postoperative intravenous fluid restriction on recovery after elective colorectal surgery. Br J Surg 93:1469-74.
5. Arkilic CF, Taguchi A, Sharma N, et al (2003). Supplemental perioperative fluid administration increases tissue oxygen pressure. Surgery 133:49-55.
6. Bennett-Guerrero E, Welsby I, Dunn TJ, et al (1999). The use of a postoperative morbidity survey to evaluate patients with prolonged hospitalization after routine, moderate-risk, elective surgery. Anesth Analg 89:514-9.
7. Mythen MG, Webb AR (1995). Perioperative plasma volume expansion reduces the incidence of gut mucosal hypoperfusion during cardiac surgery. Arch Surg 130:423-9.
8. Arieff AI (1999). Fatal postoperative pulmonary edema: pathogenesis and literature review. Chest 115: 1371-77.
9. Turnage WS, Lunn JJ (1993). Postpneumonectomy pulmonary edema. A retrospective analysis of associated variables. Chest. 103:1646-50.
10. Mathru M, Blakeman BP (1993). Don't drown the "down lung". Chest 103:1644-5.
11. Jordan S, Mitchell JA, Quinlan GJ, Goldstraw P, Evans TW. The pathogenesis of lung injury following pulmonary resection. Eur Respir J 2000; 15: 790-9
12. Patel RL, Townsend ER, Fountain SW (1992). Elective pneumonectomy: factors associated with morbidity and operative mortality. Ann Thorac Surg 54: 84-8
13. Prien T, Backhaus N, Pelster F, Pircher W, Bunte H, Lawin P (1990). Effect of intraoperative fluid administration and colloid osmotic pressure on the formation of intestinal edema during gastrointestinal surgery. J Clin Anesth 2: 317-23
14. Heughan C, Ninikoski J, Hunt TK (1972). Effect of excessive infusion of saline solution on tissue oxygen transport. Surg Gynecol Obstet 135: 257-60
15. Janvrin SB, Davies G, Greenhalgh RM (1980). Postoperative deep vein thrombosis caused by intravenous fluids during surgery. Br J Surg. 67:690-3
16. Hartmann M, Jönsson K, Zederfeldt B (1992). Effect of tissue perfusion and oxygenation on accumulation of collagen in healing wounds. Randomized study in patients after major abdominal operations. Eur J Surg 158:521-6.
17. Mutoh T, Lamm WJ, Embree LJ, Hildebrandt J, Albert RK (1992). Volume infusion produces abdominal distension, lung compression, and chest wall stiffening in pigs. J Appl Physiol 72: 575-82
18. Ratner LE, Smith GW (1993). Intraoperative fluid management. Surg Clin North Am 73: 229-41
19. Moore FD, Shires G (1967). Moderation. Ann Surg 166:300-1.
20. Alsous F, Khamiees M, Manthous CA, et al (2000). Negative fluid balance predicts survival in patients with septic shock: a retrospective pilot study. Chest 117: 1749-54.
21. Callum KG, Gray AJG, Hoile RW, et al (1999) Extremes of age: the 1999 report of the national confidential enquiry into perioperative deaths. London: National Confidential Enquiry into Perioperative Deaths.

ELIGIBILITY:
Inclusion Criteria:

* Men and women > 18 years old
* ASA I-III
* Undergoing elective general or orthopedic surgery

Exclusion Criteria:

* Emergency procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from both sexes >18 y/o, undergoing elective general or orthopedic surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Idit Matot, MD, Study Chair — Department of Anesthesia and intensive care, Tel Aviv Sourasky Medical Center; Yifat Klein, PhD, Principal Investigator — Department of Anesthesia and intensive care, Tel Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky medical center, Tel Aviv, Israel